CLINICAL TRIAL: NCT01203176
Title: Incidence of Malignant and Pre-malignant Findings in Endometrial Polyp in Asymptomatic and Symptomatic Postmenopausal Women
Brief Title: Incidence of Malignant and Premalignant Endometrial Polyp in Asymptomatic and Symptomatic Postmenopausal Women
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Arie Lissak, MD (Other)
Responsible Party: Sponsor-Investigator, Arie Lissak, MD, Head of gynecologic minimally invasive surgery unit, Carmel Medical Center., Carmel Medical Center
Organization: Carmel Medical Center (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: CMC-08-0073 CTIL
Record Dates: First submitted 2010-08-31; First posted 2010-09-16 (Estimated); Last update posted 2013-12-03 (Estimated); Status verified 2013-12

CONDITIONS: Endometrial Polyp.; Malignant and Pre-malignant Changes in the Polyp
Keywords: Endometrial polyp; Endometrial carcinoma; Endometrial hyperplasia; Postmenopausal symptomatic women; Postmenopausal asymptomatic women
MeSH Terms: conditions — Endometrial Neoplasms; Endometrial Hyperplasia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Post-menopausal symptomatic women (Active Comparator)
  Interventions: Procedure: Hysteroscopic polypectomy
- Post-menopausal asymptomatic women (Experimental)
  Interventions: Procedure: Hysteroscopic polypectomy

INTERVENTIONS:
Procedure: Hysteroscopic polypectomy — Hysteroscopy is a well established minimally invasive surgery method for diagnostic and intervention operations inside the uterine cavity. Using this method one can observe the endometrium and remove polyps.

SUMMARY:
The prevalence of endometrial polyp is 24% in the general population but is much higher in postmenopausal women. The incidence of malignant or pre-malignant findings in endometrial polyps ranges from 2 to 10% in menopausal women.

Removal of endometrial polyps in postmenopausal symptomatic women is the standard of care, same goes for asymptomatic women with risk factors for endometrial malignancy, however treatment of asymptomatic postmenopausal women with endometrial polyp but no risk factors is disputable.

In light of ambiguity in literature regarding the rate of malignant and pre-malignant findings in polyps in asymptomatic post-menopausal women, the investigators are asking to conduct a prospective study in order to evaluate and compare the incidence of malignant and pre-malignant changes in symptomatic and asymptomatic postmenopausal women with endometrial polyp

DETAILED DESCRIPTION:
Endometrial polyp is a common finding in postmenopausal women. The prevalence of endometrial polyps is 24% in the general population, but is much higher in postmenopausal in compare to premenopausal women. The incidence of malignant or pre-malignant findings in endometrial polyps ranges from 0.5 to 4.8% in the general population and from 2 to 10% in menopausal women. There is an increased risk for malignant or pre-malignant polyp in postmenopausal women and it correlates with age.

Removal of endometrial polyps in postmenopausal symptomatic (bleeding, pain, vaginal discharge) women is the standard of care, same goes for asymptomatic women with risk factors (e.g., hypertension, history of breast, ovary, endometrial or colon cancer, Tamoxifen or estrogen treatment, over-weight, no ovulation, previous endometrial hyperplasia) due to a relatively high risk for malignancy. However treatment of asymptomatic postmenopausal women endometrial polyp but no risk factors is disputable.

Article published in the recent years introduced a similar rate of involvement of malignant and pre-malignant changes in polyps removed from post-menopausal women, symptomatic and asymptomatic (3.2% versus 3.9%, respectively).

In light of ambiguity in literature regarding the rate of malignant and pre-malignant findings in polyps in asymptomatic post-menopausal women, and in light of the fact that all major studies in this field were made retrospectively, we are asking to conduct a prospective study in order to evaluate and compare the incidence of malignant and pre-malignant changes in symptomatic and asymptomatic postmenopausal women with endometrial polyp

ELIGIBILITY:
Inclusion Criteria:

1. Postmenopausal symptomatic women with Ultrasonographic or other imaging findings that correlates with endometrial polyp.
2. Postmenopausal asymptomatic women with Ultrasonographic or other imaging findings that correlates with endometrial polyp
3. Women who can read and understand and sign consent form
4. Women between 18 and 80 years of age.
5. ASA (American Society of Anesthesiologist) physical status grade 1-3

Exclusion Criteria:

1. Histological Evidence of endometrial malignancy
2. Asymptomatic woman with endometrial polyps smaller than 4 mm with no risk factors that fulfills one of the following conditions:

   * Immune depressed or terminal illness.
   * Women under anticoagulant treatment that its discontinuation, as a precondition for medical surgical intervention, could endanger their health.

Ages: 18 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1400 (Estimated)
Dates: Start 2010-09; Primary Completion 2014-08 (Estimated); Study Completion 2014-08 (Estimated)

PRIMARY OUTCOMES:
Incidence of malignant and pre-malignant changes in polyps removed from symptomatic and asymptomatic post-menopausal women | 3 years
Sonographic characteristics and histo-pathologic measures of endometrial polyp | 3 years

SECONDARY OUTCOMES:
Rate of complications during or around the operation | 3 years
Correlation between the sonographic characteristics and histopathological findings | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Arie Lissak, MD, Principal Investigator — Carmel Medical Center
Locations (1):
- Carmel Medical Center, Haifa, Israel